CLINICAL TRIAL: NCT02650622
Title: Genetic Regulators of Metabolism and Development in Children
Brief Title: Genetic and Metabolic Disease in Children
Status: Recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Ralph Deberardinis, PROFESSOR, University of Texas Southwestern Medical Center
Other Study IDs: STU 112014-001
Record Dates: First submitted 2016-01-06; First posted 2016-01-08 (Estimated); Last update posted 2025-06-26 (Actual); Status verified 2024-06

CONDITIONS: Genetic Diseases; Metabolic Diseases
Keywords: Metabolism; Genetics; Metabolomics; Genomics
MeSH Terms: conditions — Genetic Diseases, Inborn; Metabolic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — There are 3 cohorts in this study:
  Cohort 1: healthy newborns Cohort 2: healthy children aged 0-18 years old Cohort 3: Children with genetic/metabolic disorders and their families
  Blood samples will be collected from all the three cohorts for isolation of plasma for metabolomic analysis.
  In addition, DNA will be extracted from the blood samples of cohort 3 patients for genomic sequencing, and skin fibroblast cells will be collected from the proband patients in cohort 3.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Cohort 1-Newborns aged 1-2 days: No intervention will be applied specifically for this cohort. Blood samples will be collected from this cohort by piggybacking the state-mandated newborn screening test.
- Cohort 2-Children aged 0-18 years: No intervention will be applied specifically for this cohort. Blood samples will be collected from this cohort by piggybacking the blood draw of patient's standard of care.
- Cohort 3-Diseased childrens and families: Blood samples will be collected from this cohort by piggybacking the blood draw of patient's standard of care. Skin biopsy will be performed on the proband children with the agreement from parents or guardians.
  Interventions: Procedure: Skin Biopsy

INTERVENTIONS:
Procedure: Skin Biopsy — Skin biopsy will only be performed on the proband children in the cohort 3. A small piece of skin (less than 1/8'') will be removed using a local anesthetic cream and a punch, which will then be used for culture of skin cells and other laboratory tests on metabolic function.
  Groups: Cohort 3-Diseased childrens and families

SUMMARY:
This is a prospective, non-randomized, non-blinded observational study. The overarching goal is to discover new disease-associated genes in children, while establishing a specific focus on disorders where molecular characterization is most likely to lead to novel therapies. This study will merge detailed phenotypic characterization of patients presenting to the Pediatric Genetics and Metabolism Division in the Department of Pediatrics/Children's Medical Center at Dallas and collaborating clinics with Next-Generation sequencing techniques to identify disease-producing mutations. The primary objective of the study is to identify novel pathogenic mutations in children with rare Mendelian disorders. A secondary objective of the study is to establish normative ranges of a large number of metabolites from healthy newborns and older children.

DETAILED DESCRIPTION:
Discovery of genetic basis of impaired metabolism has greatly advanced treatment of patients with known metabolic diseases. However, many more genetic and metabolic disorders and their molecular causes remain to be discovered. The overall goal of this study is to discover new disease-associated genes in children, while establishing a specific focus on metabolic disorders where molecular characterization is most likely to lead to novel therapies. The primary objective is to identify novel pathogenic mutations in children with rare Mendelian disorders. The secondary objectives are: 1) Optimize methodology for metabolomic sample collection, processing and analysis; and 2) Establish normative ranges for a large number (potentially up to 1000) of metabolites in healthy newborns and older children.

Approximately one in three admissions to tertiary care pediatric hospitals results from conditions with a genetic basis. Although the majority of these conditions are rare, they collectively account for a disproportionate amount of illness and death in children. Discovery of the genetic basis of rare conditions often uncovers the pathophysiological basis of common diseases. This is particularly true for genetic diseases of impaired metabolism (inborn errors of metabolism, IEMs). There are many more genetic and metabolic disorders yet to be discovered. Of approximately 20,000 known human genes, less than one-fifth are currently associated with a disease phenotype. IEMs are a particular area of focus for us for two major reasons. First, of the several hundred known IEMs, many are already effectively treated with dietary modifications and/or medical therapy. This indicates to us that discovery of new IEM genes has great potential to produce clinically actionable insights into pathophysiology and therapeutic opportunities, ultimately leading to treatment of children that would otherwise be impossible to treat. Second, the PI of this study, Dr. Ralph DeBerardinis, is an expert in metabolomics, the practice of identifying and quantifying metabolites from biological systems. We will therefore implement research-based metabolomic profiling to the evaluation of patients with suspected IEMs or other genetic diseases. This detailed analysis will substantially increase the likelihood of identifying clinically relevant metabolic perturbations in children with growth failure, acidosis, hypoglycemia, hyperammonemia, and other abnormalities of putative genetic origin. It would also enable us to interpret mutations uncovered by clinical or research-based genomic sequencing. We believe that establishing a systematic procedure to evaluate both the metabolome and the genome in sick children will produce new insights into the genetic basis of pediatric disease, and ultimately new ways to treat these conditions.

In this study, subjects will be recruited as two populations: control and diseased. In the control population, plasma samples of healthy newborns will be acquired at the time of blood collection for state-mandated newborn screening from Parkland. We will also collect blood from healthy children from the clinics at Children's Medical Center (CMC), again piggybacking this research sample with venipuncture for clinically indicated blood collection. All plasma samples will be subjected to metabolomics to determine the healthy ranges for a large number of metabolites. This comprehensive profile of metabolites in children will be used as normative ranges to identify outlying metabolites in diseased subjects. Additionally, if suspected metabolic outliers are detected from this normal population, DNA samples extracted from the leftover packed cells or blood samples will be subjected to genomic sequencing to profile the associated gene mutations. The diseased population will be recruited from the clinics of the Pediatric Genetics and Metabolism Division in the Department of Pediatrics/CMC. Blood and DNA samples will be collected from patients for metabolomic analysis and next-generation sequencing respectively to define the metabolic abnormalities and associated gene mutations. Skin fibroblasts from patients will also be collected and used for biological validation of the metabolic effects of novel mutations, in particular by complementing diseased fibroblasts with wild-type alleles of genes mutated in the patient. If any rare Mendelian disorder is considered in a subject, blood from his/her family members will be acquired and subjected to metabolomic and genomic analyses to facilitate identification of the diseased-associated genes.

ELIGIBILITY:
Inclusion criteria of Cohort 1- Newborn:

* Subjects aged 1-2 days
* Subjects with gestational age 37-42 weeks
* Subjects with stable clinical status (admitted to normal newborn nursery)

Inclusion criteria of Cohort 2 - Older children:

• Subjects aged 0-18 years

Inclusion criteria of Cohort 3 - Diseased children:

Subjects (no age limit) with ANY phenotype as below:

* Confirmed metabolic or genetic diseases
* Suspected metabolic or genetic diseases
* Episodic metabolic decompensation (e.g. hypoglycemia, hyperammonemia, metabolic acidosis)
* Developmental regression
* Major congenital malformation
* Other unexplained symptoms of potential genetic origin

Exclusion criteria of Cohort 1 - Newborn:

* Subjects with gestational age <37 weeks or >42 weeks
* Subjects with overt signs of metabolic dysfunction, distress or genetic diseases including hypoglycemia, hyperglycemia, sepsis/shock, hypoxemia, or major congenital malformation
* Subjects with mothers whose pregnancies were complicated by gestational diabetes, gestational hyperglycemia, gestational hypertension, preeclampsia, or any other major disorders.

Exclusion criteria of Cohort 2 - Older children:

* Subjects with confirmed metabolic or genetic diseases
* Subjects with suspected metabolic or genetic diseases
* Subjects with episodic metabolic decompensation (e.g. hypoglycemia, hyperammonemia, metabolic acidosis)
* Subjects with developmental regression
* Subjects with major congenital malformation

Exclusion criteria of Cohort 3 - Diseased children No.

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Two populations will be enrolled in this study, control and diseased. Healthy newborns and older children will be recruited into the control population from Parkland Postpartum units and Children's Medical Center (CMC), respectively. The diseased population will be recruited from the clinics of the Pediatric Genetics and Metabolism Division in the Department of Pediatrics of CMC.
Sampling Method: Non-Probability Sample
Enrollment: 1550 (Estimated)
Dates: Start 2015-06 (Actual); Primary Completion 2030-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Perform metabolomic profiling and exome sequencing in children with presumed genetic and metabolic diseases | 3-4 years
  The Levels of the metabolites that can be detected in the plasma from the enrolled children will be measured by mass-spectrometry technique.The DNA samples will be extracted from the blood samples of diseased children and then subjected to exome sequencing to identify gene mutations.

SECONDARY OUTCOMES:
Perform metabolomic profiling in healthy children | 3-4 years
  The Levels of the metabolites will be measured by by mass-spectrometry technique in the plasma samples from enrolled healthy children.

OTHER OUTCOMES:
Establish a specimen repository of healthy and diseased children | 3 years
  Blood samples and derived plasma and DNA samples, and patient fibroblast cell lines will be de-identified and stored in research laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: Ralph J DeBerardinis, MD, PhD, Principal Investigator — UT Southwestern Medical Center, Children's Medical Center at Dallas
Locations (1):
- Children's Medical Center at Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Scriver CR, Neal JL, Saginur R, Clow A. The frequency of genetic disease and congenital malformation among patients in a pediatric hospital. Can Med Assoc J. 1973 May 5;108(9):1111-5. PMID 4704890
- [Background] Ng SB, Buckingham KJ, Lee C, Bigham AW, Tabor HK, Dent KM, Huff CD, Shannon PT, Jabs EW, Nickerson DA, Shendure J, Bamshad MJ. Exome sequencing identifies the cause of a mendelian disorder. Nat Genet. 2010 Jan;42(1):30-5. doi: 10.1038/ng.499. Epub 2009 Nov 13. PMID 19915526